CLINICAL TRIAL: NCT01861600
Title: Stool Composition and Stool Characteristics in Healthy Term Infants Fed Human Milk or Infant Formulas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9055A1-3001
Record Dates: First submitted 2013-04-17; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Stool Composition
Keywords: Stool composition
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Experimental (EF) 1 (Experimental): For 8 weeks, infants will consume ad libitum per day S-26 Gold EF1
  Interventions: Other: S-26 Gold EF1
- Standard Formula (Active Comparator): For 8 weeks, infants will consume ad libitum per day. S-26 Gold
  Interventions: Other: S-26 Gold
- Experimental 2 (EF2) S-26 Gold (Experimental): For 8 weeks, infants will consume ad libitum per day. S-26 Gold EF2
  Interventions: Other: S-26 Gold EF2
- Human milk (HM) (Other): For 8 weeks, infants will consume ad libitum per day. Human Milk
  Interventions: Other: Human Milk
- Experimental formula (EF) 3 (Experimental): For 8 weeks, infants will consume ad libitum per day. S-26 Gold EF3
  Interventions: Other: S-26 Gold EF3

INTERVENTIONS:
Other: S-26 Gold — (13.4 g/L protein) with 100% Fat Blend A
  Arms: Standard Formula
Other: S-26 Gold EF1 — (13.4 g/L protein) with 60% Fat Blend A and 40% Betapol fat blend
  Arms: Experimental (EF) 1
Other: S-26 Gold EF2 — (13.4 g/L protein) with 60% Fat Blend A and 40% Betapol fat blend, and supplemented with 3.0 g/L oligofructose
  Arms: Experimental 2 (EF2) S-26 Gold
Other: S-26 Gold EF3 — (13.4 g/L protein) with 60% Fat Blend A and 40% Betapol fat blend, and supplemented with 5.0 g/L oligofructose
  Arms: Experimental formula (EF) 3
Other: Human Milk — Human Milk
  Arms: Human milk (HM)

SUMMARY:
The primary efficacy objective was to determine and compare stool composition (stool soap and non-soap fatty acids, total fatty acids, minerals, and other stool constituents) among the feeding groups.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of term infant formula containing high 2-palmitic vegetable oil on stool composition and characteristics and to investigate the effect of both high 2-palmitic vegetable oil and oligofructose in infant formula on stool softness and bacteria. Because some studies demonstrate the benefit of high concentrations of a non-digestible carbohydrate in the formula, we will study 2 concentrations of added oligofructose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, term (no less than 37 weeks, 0 days and no greater than 42 weeks, 0 days) singleton infants, between 7 days and 14 day post natal age
2. Weight for age ≥5th percentile according to Filipino growth tables/charts.
3. HM infants were exclusively consuming and tolerating HM
4. Mother must have made the decision to continue to exclusively breastfeed.
5. Formula-fed infants were exclusively consuming and tolerating a cow's milk infant formula
6. Parent/guardian must have previously made the decision to continue to exclusively formula feed

Exclusion Criteria:

1. Infants who are receiving any amount of supplemental HM with infant formula feeding or visa versa
2. Infants who are receiving any infant formula containing pro- or prebiotics
3. Family history of siblings with documented cow's milk protein intolerance/allergy
4. Conditions requiring infant feedings other than those specified in the protocol
5. Major congenital malformations (e.g. cleft palate, hemangiomas, extremity malformation)
6. Suspected or documented systemic or congenital infections (e.g. human immunodeficiency virus, cytomegalovirus)
7. Evidence of significant cardiac, respiratory, endocrinologic, hematologic, gastrointestinal, or other systemic diseases
8. Infants who have received any experimental treatment, participated in any other clinical trial, or received any other investigational intervention unrelated to this trial, prior to enrollment
9. Infants of any ancillary personnel connected with the study or the infants of first and second-degree relatives (parents, brothers, sisters, children, or grandchildren) of ancillary personnel
10. Presently receiving or have received any medication(s) which are known or suspected to affect fat digestion, absorption and/or metabolism (e.g., pancreatic enzymes), any vitamin and/or mineral supplements which contain calcium, all antibiotics and antifungal medications (except topical), suppositories, bismuth-containing medications, herbal supplements, or medications which may neutralize or suppress gastric acid secretion
11. HM-fed infants whose mothers are presently receiving or have received any antibiotics or antifungal medications (except topical), post partum

Ages: 7 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Stool Composition in Healthy Term Infants Fed Human Milk or Infant Formulas | 8 weeks
  stool composition: stool soap and non-soap fatty acids, total fatty acids, minerals, and other stool constituents

SECONDARY OUTCOMES:
Stool Characteristics in Healthy Term Infants Fed Human Milk or Infant Formulas | 8 weeks
  Determinations of fecal flora as well as fecal pH, sIgA concentrations and SCFA concentrations in a subset of subjects.

OTHER OUTCOMES:
Safety evaluation | 10 weeks
  evaluation of adverse events
Growth evaluation | 8 weeks
  Anthropometric measurements

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario Zeta Capeding, MD, Principal Investigator — JRF Health Center Complex, Muntinlupa City, Philippines
Locations (1):
- Asian Hospital and Medical Center, Metro Manila, Alabang, Philippines

REFERENCES:
- [Derived] Yao M, Lien EL, Capeding MR, Fitzgerald M, Ramanujam K, Yuhas R, Northington R, Lebumfacil J, Wang L, DeRusso PA. Effects of term infant formulas containing high sn-2 palmitate with and without oligofructose on stool composition, stool characteristics, and bifidogenicity. J Pediatr Gastroenterol Nutr. 2014 Oct;59(4):440-8. doi: 10.1097/MPG.0000000000000443. PMID 24840511